CLINICAL TRIAL: NCT04324775
Title: Comparison of Acute Effect of Manual Lymph Drainage and Swedish Massage on Muscle Fascia Stiffness Applied After Exercise in Healthy Young Women
Brief Title: Comparison of Acute Effect of Different Manual Techniques on Muscle Fascia Stiffness
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2019.968
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-01

CONDITIONS: Manual Lymphatic Drainage; Swedish Massage; Muscle Fascia Stiffness
Keywords: MLD, massage, fascia, stiffness
MeSH Terms: conditions — Leukodystrophy, Metachromatic | interventions — Exercise; Manual Lymphatic Drainage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Exercise+Manual Lymphatic Drainage
  Interventions: Other: Exercise + Manual Lymphatic Drainage
- Group 2: Exercise+Swedish Massage
  Interventions: Other: Exercise + Swedish massage

INTERVENTIONS:
Other: Exercise + Manual Lymphatic Drainage — Quadriceps exercises with weight of 75%1 Max repetition and 8 repetionX3 sets Following exercises, manual lymphatic drainage applied to rectus femoris for 5 minutes
  Groups: Group 1
Other: Exercise + Swedish massage — Quadriceps exercises with weight of 75%1 Max repetition and 8 repetionX3 sets Following exercises, swedish massage applied to rectus femoris for 5 minutes
  Groups: Group 2

SUMMARY:
There are studies investigating the effect of different massage methods on muscle fascia stiffness but the results do not support each other. In addition, there is no study to investigate the effect of MLD on muscle fascia stiffness. The aim of this study is to determine the acute effect of MLD and classical (Swedish) massage (KM) on muscle fascia stiffness after exercise.

ELIGIBILITY:
Inclusion Criteria:

* Being health and woman
* No systemic problem preventing exercise
* Having sufficient level of perception to perceive commands
* BMI≤25

Exclusion Criteria:

* Having a history of injury and surgery through the Quadriceps femoris muscle in the last three months
* Having a disease that will affect myofascial structure features
* Having a disease that will affect normal body temperature
* Chronic pain in Quadriceps femoris muscle that has been going on for the last three months.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Volunteer woman healthy student between the ages of 18-25 with a subcutaneous fold thickness of the quadriceps muscle between 5 mm and 15 mm.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-04-15 (Estimated); Study Completion 2020-04-20 (Estimated)

PRIMARY OUTCOMES:
Measurement of skin temperature | Change from Baseline skin temperature at following exercises, at following MLD/SM application and at 10 minutes after the exercise
  For thermal imaging, a 120-9-90 pixel resolution FLIR E5 camera thermal camera (FLIR Systems AB, Sweden) will be used, and Color Palette iron will be selected to display images. The video will be taken from a distance of 1 m at a speed of 8 photos / s.
Evaluation of the mechanical properties of the muscle-1 | Change from Baseline mechanical properties at following exercises, at following MLD/SM application and at 10 minutes after the exercise
  Viscoelastic stiffness [N/m] will be measured in MyotonPro 3 (MYO, Tallin, Estonia).
Evaluation of the mechanical properties of the muscle-2 | Oscillation frequency (Hz) will be measured in MyotonPro 3 (MYO, Tallin, Estonia)
  Change from Baseline mechanical properties at following exercises, at following MLD/SM application and at 10 minutes after the exercise
Evaluation of the mechanical properties of the muscle-3 | Change from Baseline mechanical properties at following exercises, at following MLD/SM application and at 10 minutes after the exercise
  Mechanical stiffness (N/m) will be measured in MyotonPro 3 (MYO, Tallin, Estonia).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakar Y, Coknaz H, Karli U, Semsek O, Serin E, Pala OO. Effect of manual lymph drainage on removal of blood lactate after submaximal exercise. J Phys Ther Sci. 2015 Nov;27(11):3387-91. doi: 10.1589/jpts.27.3387. Epub 2015 Nov 30. PMID 26696704
- [Background] Kong PW, Chua YH, Kawabata M, Burns SF, Cai C. Effect of Post-Exercise Massage on Passive Muscle Stiffness Measured Using Myotonometry - A Double-Blind Study. J Sports Sci Med. 2018 Nov 20;17(4):599-606. eCollection 2018 Dec. PMID 30479528
- [Background] Ogai R, Yamane M, Matsumoto T, Kosaka M. Effects of petrissage massage on fatigue and exercise performance following intensive cycle pedalling. Br J Sports Med. 2008 Oct;42(10):834-8. doi: 10.1136/bjsm.2007.044396. Epub 2008 Apr 2. PMID 18385196
- [Result] Eriksson Crommert M, Lacourpaille L, Heales LJ, Tucker K, Hug F. Massage induces an immediate, albeit short-term, reduction in muscle stiffness. Scand J Med Sci Sports. 2015 Oct;25(5):e490-6. doi: 10.1111/sms.12341. Epub 2014 Dec 8. PMID 25487283